CLINICAL TRIAL: NCT01770392
Title: Relative Bioavailability of a Single Oral Dose of Nintedanib Given Alone and in Combination With Multiple Oral Doses of Rifampicin in Healthy Male Volunteers (an Open-label, Two-period, Fixed Sequence Phase I Trial)
Brief Title: Relative Bioavailability of a Single Dose of Nintedanib Given Alone and in Combination With Multiple Doses of Rifampicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.162; 2012-002507-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib; Rifampin

ARMS (2):
- Test (Active Comparator): multiple doses of Rifampicin + single dose of Nintedanib
  Interventions: Drug: Rifampicin; Drug: Nintedanib
- Reference (Experimental): single dose of Nintedanib
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — single dose administration
  Arms: Reference
Drug: Rifampicin — single dose once daily for 7 days
  Arms: Test
Drug: Nintedanib — single dose administration
  Arms: Test

SUMMARY:
To investigate the effect of the P-gp inducer rifampicin on the pharmacokinetic parameters of nintedanib

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1199.162.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Luedtke D, Marzin K, Jungnik A, von Wangenheim U, Dallinger C. Effects of Ketoconazole and Rifampicin on the Pharmacokinetics of Nintedanib in Healthy Subjects. Eur J Drug Metab Pharmacokinet. 2018 Oct;43(5):533-541. doi: 10.1007/s13318-018-0467-9. PMID 29500603

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This was an open-label, two-period, fixed-sequence trial. During the first period 150 mg of nintedanib was administered orally in form of a soft gelatine capsule. In the second period, a single dose of 600 mg of rifampicin was administered orally via film-coated tablet every day for a week, then a single dose of nintedanib was administered. The administrations of nintedanib were separated by a washout period of at least 14 days.
Period: Nintedanib
Arm/Group | Overall Study
Started | 26
Completed | 26
Not Completed | 0
Period: Washout Period of at Least 14 Days
Arm/Group | Overall Study
Started | 26
Completed | 25
Not Completed | 1
Not completed — Adverse Event | 1
Period: Nintedanib+ Rifampicin
Arm/Group | Overall Study
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consists of all subjects who took at least one dose of study medication.
Arm/Group | Overall Study
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞ represents the Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity.
  For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1.5 hour (h) before the first drug administration and 0.5h, 1h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h and 72h after administration of nintedanib
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Nintedanib: 150 mg of nintedanib was given as a single dose on Day 1.
- Nintedanib + Rifampicin: 600 mg rifampicin was given every evening from Day -7 to Day -1, followed by a single dose of 150 mg nintedanib in the morning of Day 1.
Arm/Group | Nintedanib | Nintedanib + Rifampicin
Number analyzed (Participants) | 26 | 25
ng*h/mL | 183 (36.1) | 89.4 (36.8)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Rifampicin; Test type: Superiority or Other; p = 1.0000, ANOVA — p-value for ratio outside interval 0.8 - 1.25; The model includes fixed effect for treatment and effect "subjects" was considered as random; Geometric Mean Ratio in percentage = 50.12, 90% CI 2-sided [47.155 to 53.275], Standard Deviation 12.7 — The standard deviation is actually the geometric coefficient of variation (in %). The ratio has been calculated as (nintedanib+ rifampicin) divided by nintedanib (in %)

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Cmax represents the maximum concentration of nintedanib in plasma. For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib | Nintedanib + Rifampicin
Number analyzed (Participants) | 26 | 25
ng/mL | 22.1 (51.8) | 12.8 (43.4)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Rifampicin; Test type: Superiority or Other; p = 1.0000, ANOVA — p-value for ratio outside interval 0.8 - 1.25; The model includes fixed effect for treatment and effect "subjects" was considered as random; Geometric Mean Ratio in percentage = 59.76, 90% CI 2-sided [53.829 to 66.348], Standard Deviation 21.9 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Curve From 0 to the Last Quantifiable Concentration (AUC0-tz)
Description: AUC0-tz represents the area under the plasma concentration-time curve of nintedanib from 0 to the last quantifiable analyte plasma concentration.
  For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib | Nintedanib + Rifampicin
Number analyzed (Participants) | 26 | 25
ng*h/mL | 173 (36.9) | 84.1 (38.1)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Rifampicin; Test type: Superiority or Other; p = 1.0000, ANOVA — p-value for ratio outside interval 0.8 - 1.25; The model includes fixed effect for treatment and effect "subjects" was considered as random; Geometric Mean Ratio in percentage = 49.98, 90% CI 2-sided [46.886 to 53.286], Standard Deviation 13.3 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first trial drug administration until up to 14 days after last trial drug administration, up to 28 days
Groups:
- Washout Period: washout period of at least 14 days between the administrations of nintedanib. During this period no trial drug was administered
- Rifampicin: 600 mg rifampicin was given every evening from Day -7 to Day -1
Arm/Group | Nintedanib | Washout Period | Rifampicin | Nintedanib + Rifampicin
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/26 | 2/26 | 25/25 | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=26) | Washout Period (N=26) | Rifampicin (N=25) | Nintedanib + Rifampicin (N=25)
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1 | 3
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 25 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights